CLINICAL TRIAL: NCT01304914
Title: Prospective, Community-based, Longitudinal Dynamic Birth Cohort Study of Respiratory and Gastrointestinal Pathogen Identification in Brisbane Infants.
Brief Title: Observational Research in Childhood Infectious Diseases Study
Acronym: ORChID
Status: Completed | Type: Observational
Sponsor: The University of Queensland (Other)
Collaborators: Royal Brisbane and Women's Hospital (Other Government)
Responsible Party: Principal Investigator, Dr Stephen Lambert, Senior Research Fellow, The University of Queensland
Other Study IDs: HREC10/QRCH16
Record Dates: First submitted 2011-02-25; First posted 2011-02-28 (Estimated); Last update posted 2016-03-31 (Estimated); Status verified 2016-03

CONDITIONS: Respiratory Tract Infections; Gastrointestinal Infections
Keywords: Respiratory tract infections; Gastrointestinal tract infections; Pediatrics; Specimen collection
MeSH Terms: conditions — Respiratory Tract Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Parent-collected anterior-nasal swabs Nappy swabs
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Healthy, term-delivered babies

SUMMARY:
In this study, the investigator will be approaching pregnant women to undertake 2 years of weekly respiratory and nappy specimen collection from their healthy new born infant. These specimens will be mailed to the Queensland Paediatric Infectious Diseases (Qpid) Laboratory where they will be stored and batched tested for viruses and bacteria. As well as this, parents will keep a simple daily symptom diary for their child, allowing us to match detection of viruses and bacteria to periods when the study child did or did not have symptoms. This will help our understanding of what finding these viruses and bacteria in specimens from children really means.

DETAILED DESCRIPTION:
This will be a prospective, community-based longitudinal birth cohort study of respiratory and gastrointestinal pathogen detection in Brisbane infants. The enrollment target of 138 children will take 2 years to achieve, each child will be followed until their second birthday, and a final year will be required for specimen and data analysis; for a total duration of the study of 5 years.

Women are to be recruited antenatally over a period of two years from study commencement (mid-2010). These hospitals serve communities from the north of Brisbane, a city of almost 2 million people, and every year each has roughly 5,200 (RBWH) and 1,700 (North West) annual deliveries respectively. The investigators will follow 138 infants from birth until their second birthday. Where a family drops out of the study or is lost to follow-up, they will be replaced to maintain overall person-time for the study.

The progressive 2 year recruitment plan allows for seasonal and year-to-year variation in respiratory virus activity. Eligible infants will be healthy term babies without conditions that predispose to more frequent or severe infectious episodes.

Parents will keep a simple, daily, infection symptom diary, completed using tick boxes and numbers, which the investigators will request be returned on a 4-weekly basis. A similar diary was used for a 12-month cohort study conducted in Melbourne (2003-2004) with excellent return rate and acceptability by study families.

Study families are to be contacted monthly by their preferred method of communication (telephone, SMS, or email) to encourage continued performance of study tasks and answer study related questions.

Parents will be asked to identify acute respiratory illness (ARI) and acute gastroenteritis (AGE) in study children. These are defined as:

* ARI: presence of at least one yellow OR at least two blue symptoms on a single day; and
* AGE: three or more watery or looser-than-normal stools OR vomiting on a single day.

When an ARI or AGE occur, parents will be asked to complete an impact diary for the duration of illness. Parents will be asked to contact us in the event of hospitalisation due to any cause. Parents will be asked to provide consent for hospital/GP release of information to allow study staff to collect details of episodes of care.

Cord blood will also be collected at birth and stored for later identification of pathogen-specific antibodies and immune mediators linked to disease susceptibility. A respiratory and stool swab will be collected from study neonates within one day of birth. At this visit, the investigators will collect a respiratory swab from the parent/s of the child - this will allow us to compare presence of pathogens in the neonate and parents, and will be the only time parents will be swabbed. Parents will be trained in the process of collecting the study swabs at this visit. All material and instructions required for this process will be provided to parents at no cost. Telephone and visiting support to assist and guide specimen collection will be available for study parents at all stages during the study.

Parents will be asked to routinely collect two specimens on the same day of the week as the initial visit, weekly until the end of the study. The specimens are:

* a combined anterior nares swab, collected from both nostrils using a single, rayon-budded swab. The swab comes with its own transport tube containing a VTM-soaked sponge in the base. The completed swab is placed in the transport tube and the VTM sponge is squeezed to bath the swab; and
* a stool swab from a dirty nappy, collected and handled using the swab similar to the anterior nares swab.

Both swabs are mailed back to Qpid Laboratory as soon as possible after collection, using pre-addressed, reply post, padded envelopes.

All specimens will be batch tested for a variety of pathogens using validated PCR methods developed at Qpid. Samples from children with ARI or AGE for whom a known agent cannot be identified, will be made available for further investigations for the presence of as yet unidentified viruses.

ELIGIBILITY:
Inclusion Criteria:

* pregnant women expecting to deliver a healthy, term baby
* written informed consent from pregnant woman who is available for telephone contact for the duration of the study, and not planning to move out of the study area
* parent willing to collect a weekly anterior nasal specimen and stool (nappy) specimen from the study child and return to study site via mail
* parent or guardian with sufficient English language skills to complete study diaries and perform study tasks as required

Exclusion Criteria:

* children born before 36 weeks
* children with chronic pulmonary or cardiovascular disorders
* children with chronic metabolic disorders (such as, but not limited to, diabetes mellitus, renal dysfunction, haemoglobinopathies)
* children with immune system disorders (such as HIV/AIDS or receiving immune system suppressing medications)
* children with other chronic illnesses whose enrollment is deemed by the investigators to make it inappropriate to enroll them onto, or to continue in, the study

Max Age: 7 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Healthy, term-delivered babies
Sampling Method: Non-Probability Sample
Enrollment: 165 (Actual)
Dates: Start 2010-08; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Acute respiratory illness (ARIs) and acute gastrointestinal (AGE) illness rates per 10,000 child-days in healthy children in the first two years of life | Two years
  This measure will be calculated using counts of ARIs and AGE in study children during the first two years of life as the numerator, and person-time in child-months on the study as the denominator.

SECONDARY OUTCOMES:
Pathogen-specific rate of episodes of ARI and AGE per 10,000 child-days in healthy children in the first two years of life | 2 years
  Viral and bacterial testing will allow to calculate pathogen-specific rates: This measure will be calculated using counts of pathogen-specific ARIs and AGE in study children during the first two years of life as the numerator, and person-time in child-months on the study as the denominator.
Detection of novel pathogens in healthy children in the first 2 years of life. | 2 years
  A subset of samples collected during this study will be used to attempt to identify previously undetected pathogens in children, through microarray technology and random primer PCR testing.

CONTACTS AND LOCATIONS:
Overall Officials: Keith Grimwood, MD, Principal Investigator — The University of Queensland; Theo P Sloots, PhD, Principal Investigator — The University of Queensland; Michael D Nissen, FRACP, Principal Investigator — The University of Queensland; Stephen B Lambert, PhD, Principal Investigator — The University of Queensland
Locations (2):
- Australia (2):
  - Royal Brisbane and Women's Hospital, Brisbane, Queensland
  - Northwest Private Hospital, Everton Park, Queensland

REFERENCES:
- [Derived] Saha S, Fozzard N, Grimwood K, Lambert SB, Ware RS. The Ages When Healthy Children Are First Colonized by Three Common Potentially Pathogenic Bacteria: A Birth Cohort Study. Pediatr Infect Dis J. 2025 Apr 3;44(9):907-909. doi: 10.1097/INF.0000000000004798. PMID 40208931
- [Derived] El-Heneidy A, Grimwood K, Mihala G, Lambert S, Ware RS. Epidemiology of Norovirus in the First 2 Years of Life in an Australian Community-based Birth Cohort. Pediatr Infect Dis J. 2022 Nov 1;41(11):878-884. doi: 10.1097/INF.0000000000003667. Epub 2022 Oct 11. PMID 36223234
- [Derived] Wang CYT, Ware RS, Lambert SB, Mhango LP, Tozer S, Day R, Grimwood K, Bialasiewicz S. Parechovirus A Infections in Healthy Australian Children During the First 2 Years of Life: A Community-based Longitudinal Birth Cohort Study. Clin Infect Dis. 2020 Jun 24;71(1):116-127. doi: 10.1093/cid/ciz761. PMID 31406985
- [Derived] Ye S, Whiley DM, Ware RS, Kirkwood CD, Lambert SB, Grimwood K. Multivalent Rotavirus Vaccine and Wild-type Rotavirus Strain Shedding in Australian Infants: A Birth Cohort Study. Clin Infect Dis. 2018 Apr 17;66(9):1411-1418. doi: 10.1093/cid/cix1022. PMID 29149283
- [Derived] Sarna M, Alsaleh A, Lambert SB, Ware RS, Mhango LP, Mackay IM, Whiley DM, Sloots TP, Grimwood K. Respiratory Viruses in Neonates: A Prospective, Community-based Birth Cohort Study. Pediatr Infect Dis J. 2016 Dec;35(12):1355-1357. doi: 10.1097/INF.0000000000001316. PMID 27580059
- [Derived] Lambert SB, Ware RS, Cook AL, Maguire FA, Whiley DM, Bialasiewicz S, Mackay IM, Wang D, Sloots TP, Nissen MD, Grimwood K. Observational Research in Childhood Infectious Diseases (ORChID): a dynamic birth cohort study. BMJ Open. 2012 Oct 31;2(6):e002134. doi: 10.1136/bmjopen-2012-002134. Print 2012. PMID 23117571